CLINICAL TRIAL: NCT04932850
Title: COVID-19: A Phase I Dose-escalation Study to Evaluate the Safety and Pharmacokinetics of Anti-SARS-CoV-2 Monoclonal Antibody MAD0004J08 in Healthy Adults.
Brief Title: Study to Evaluate the Safety and Concentrations of Monoclonal Antibody Against Virus That Causes COVID-19 Disease.
Acronym: MAD0004J08
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Toscana Life Sciences Sviluppo s.r.l. (Industry)
Collaborators: Cross Research S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A0001A; 2020-005469-15 (EudraCT Number)
Record Dates: First submitted 2021-06-15; First posted 2021-06-21 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: COVID-19 Virus Disease
Keywords: COVID-19 Pandemic; SARS-CoV-2 Infection; SARS-CoV-2 Monoclonal Antibody
MeSH Terms: conditions — COVID-19 | interventions — MAD0004J08

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Identical kits for active and placebo will be provided.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): 3 active cohorts are involved into study: Cohort 1 (48 mg), Cohort 2 (100 mg) and Cohort 3 (400 mg).
  Each cohort is composed of two groups. The subjects enrolled in the first group of each cohort (groups 1, 3 and 5 for Cohorts 1, 2 and 3, respectively) will be sentinel subjects and will be treated one at the time at 48 h intervals in order to evaluate possible treatment-related adverse events.
  Interventions: Biological: MAD0004J08
- Placebo (Placebo Comparator): Placebo will be administered to 2 subjects for each cohort.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MAD0004J08 — Human mAb 100 mg / 2.5 mL solution for injection
  Arms: Active
Other: Placebo — Placebo matching to MAD0004J08 2.5 mL solution for injection
  Arms: Placebo

SUMMARY:
A Phase I dose-escalation study to test a new monoclonal antibody (called MAD0004J08) against severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), the virus that causes COVID-19 disease. The study aims to evaluate the safety and pharmacokinetics (distribution and elimination) of anti-SARSCoV-2 monoclonal antibody in healthy adults.

The primary objective of the study is to evaluate the safety of anti-SARSCoV-2 monoclonal antibody (that is the appearance of adverse events), the pharmacokinetics (how MAD0004J08 is distributed and eliminated by human body), the generation of anti-drug antibodies (ADAs) (that is the possible production of antibodies against the drug, which could invalidate it efficacy) and finally the ability of MAD0004J08 to neutralize SARSCoV-2. Furthermore a blood sample would be used to evaluate a kit (DIESSE kit), developed by Toscana Life Sciences, able to detect the administered drug. This kit is not used to evaluate study paramethers.

30 subjects, that should respect the Inclusion/Exclusion criteria, will be enrolled.

About 12 visits will be performed during the study, study duration will be about 6 months.

Subjects will be distributed into 3 Cohorts, each of them divided into 2 groups that would receive MAD0004J08 (Dose 1 = 48 mg, Dose 2 = 100 mg or Dose 3 = 400 mg) or placebo. Administration occurs as intramuscular injection (single injection for Cohort 1 and Cohort 2 and, two injections for Cohort 3) .

DETAILED DESCRIPTION:
A Phase I dose-escalation study to evaluate the safety and pharmacokinetics of anti-SARSCoV- 2 monoclonal antibody MAD0004J08 in healthy adults.

Two Italian clinical sites are involved in the study. It is a first-in-human, single-dose, dose-escalation, double-blind, placebo-controlled, randomised, safety and pharmacokinetics study.

Three single ascending doses (48 mg, 100 mg and 400 mg) and placebo will be administered by intramuscular injection to three study cohorts (10 subjects/cohort) as single doses, in the morning of day 1.

There are 5 sentinel subjects for each Cohort, they will be treated one at the time at 48 h distance (after evaluation of any possible treatment related adverse event).

Active treatment and placebo will be assigned within each cohort and group according to the study randomisation list.

Go/No-go decision on escalation from Cohort 1 to Cohort 2 and from Cohort 2 to Cohort 3 will be taken after evaluation of Cohort 1/Cohort 2 safety data up to 48 h post-dose by an independent Data Safety Monitoring Board.

The primary objective of the study is to evaluate the safety of three single dose levels of MAD0004J08 in healthy subjects.

Secondary objectives are to evaluate the pharmacokinetics of MAD0004J08, potency in terms of serum neutralisation power and immunogenicity in terms of generation of anti-drug antibodies (ADAs) after single dose of 48 mg, 100 mg and 400 mg.

The following procedures will be performed:

Visit 1 - Screening Day -21 / Day -2

* Explanation to the subject of study aims, procedures and possible risks
* Informed consent signature
* Screening number assignment (as S001, S002, etc.)
* Demographic data and life style recording
* Medical history
* Previous/concomitant medications
* Physical examination (including body weight, height)
* Vital signs (blood pressure, heart rate, body temperature)
* 12-lead Electrocardiogram (ECG)
* SARS-CoV-2 serology test
* Laboratory analyses: haematology, blood chemistry, urinalysis, serum virology, coagulation, ferritin
* Drug of abuse test
* Urinary pregnancy test (women)
* SARS-CoV-2 Real-Time Quantitative Reverse Transcription PCR (qRT-PCR) in the 72 h before day 1 (could be performed on day -3 or day-2 or day -1)
* Adverse event monitoring
* Inclusion/exclusion criteria evaluation
* Eligibility evaluation Visit 2 - Day -1
* SARS-CoV-2 qRT-PCR in the 72 h before treatment. On day -1 either test performance, or result check if already performed on day -3 or day -2
* Drug of abuse test
* Inclusion/exclusion criteria evaluation
* Check of AEs and concomitant medications
* Vital signs (blood pressure, heart rate, body temperature)
* Physical examination
* Eligibility evaluation Visit 3 - Day 1
* Urine pregnancy test (women)
* Inclusion/exclusion criteria evaluation, eligibility evaluation, and randomisation
* 12-lead ECG
* Dispensation of 2 diaries to the subject (diary 1 to report solicited adverse events from day 1 to day 8, diary 2 to report all unsolicited adverse events and concomitant medication from day 1 to month 1)
* Laboratory analyses: haematology, coagulation, blood chemistry, urinalysis, SARS-CoV-2 serology test - baseline
* Blood sample collection for pharmacokinetic analysis at predose (0) and 1h, 2h, 3h, 4h, 6h, 8h, 12h post-dose
* Blood sample collection for ADA analysis at pre-dose (0)
* Blood sample collection for serum neutralising power test at pre-dose (0)
* Blood sample collection for DIESSE Elisa kit characterisation at pre-dose (0)
* Vital signs (blood pressure, heart rate, body temperature) measurement at pre-dose (0), 2h post-dose and 12 h post-dose
* Investigational product administration (active or placebo according to study Cohort, Group and randomisation)
* Adverse events monitoring
* Injection site reactions check
* Concomitant medications check Visit 4 - Day 2
* Physical examination
* Vital signs (blood pressure, heart rate, body temperature) measurement at 24 h post-dose
* Blood sample collection for pharmacokinetic analysis at 24h post-dose
* Adverse events monitoring
* Injection site reactions check
* Diary 1 and diary 2 check
* Concomitant medications check
* Laboratory analyses: haematology, blood chemistry, coagulation, urinalysis, SARS-CoV-2 serology test at 24 h post-dose
* 12-lead ECG at 24 h post-dose Visit 5 - Day 3
* Vital signs (blood pressure, heart rate, body temperature) measurement at 48 h post-dose
* Blood sample collection for pharmacokinetic analysis at 48h post-dose
* Blood sample collection for serum neutralising power test at 48h post-dose
* Blood sample collection for DIESSE Elisa kit characterisation at 48 h post-dose
* Adverse events monitoring
* Injection site reactions check
* Diary 1 and diary 2 check
* Concomitant medications check
* Laboratory analyses: haematology, blood chemistry, coagulation, urinalysis, SARS-CoV-2 serology test - at 48 h post-dose
* Physical examination Visits 6 / Week 1 / Day 8 and Visit 7 / Week 2 / Day 15±2
* Physical examination
* Vital signs (blood pressure, heart rate, body temperature) measurement
* Blood sample collection for pharmacokinetic analysis
* Blood sample collection for ADA analysis
* Blood sample collection for serum neutralising power test on day 8 only
* Blood sample collection for DIESSE Elisa kit characterisation on day 8 only
* Adverse events monitoring
* Concomitant medications check
* Laboratory analyses: haematology, blood chemistry, coagulation, urinalysis, SARS-CoV-2 serology test
* Diary 1 check - day 8 only
* Diary 2 check - day 8 and day 15
* Subjects' diary 1 return - day 8 only Visit 8 Week 3 Day 22±2
* Physical examination
* Vital signs (blood pressure, heart rate, body temperature)
* Blood sample collection for pharmacokinetic analysis
* Adverse events monitoring
* Diary 2 check
* Concomitant medications check
* Laboratory analyses: haematology, blood chemistry, coagulation, urinalysis, SARS-CoV-2 serology test Visit 9 - 1 month Day 30±3
* Physical examination
* Vital signs (blood pressure, heart rate, body temperature) measurement
* Blood sample collection for pharmacokinetic analysis
* Blood sample collection for ADA analysis
* Blood sample collection for serum neutralising power test
* Blood sample collection for DIESSE Elisa kit characterisation
* Adverse events monitoring
* Diary 2 check
* Concomitant medications check
* Laboratory analyses: haematology, blood chemistry, coagulation, urinalysis, SARS-CoV-2 serology test
* Urine pregnancy test (women)
* Subjects' diary 2 return Visit 10 - 2 months Day 60±4
* Physical examination
* Vital signs (blood pressure, heart rate, body temperature) measurement
* Blood sample collection for pharmacokinetic analysis
* Adverse events monitoring
* Concomitant medications check
* Laboratory analyses: haematology, blood chemistry, coagulation, urinalysis, SARS-CoV-2 serology test
* Urine pregnancy test (women) Visit 11 - 4 months Day 120±4 days
* Physical examination
* Vital signs (blood pressure, heart rate, body temperature) measurement
* Blood sample collection for pharmacokinetic analysis
* Blood sample collection for ADA
* Blood sample collection for serum neutralising power test
* Blood sample collection for DIESSE Elisa kit characterisation
* Adverse events monitoring
* Concomitant medications check
* Laboratory analyses: haematology, blood chemistry, coagulation, urinalysis, SARS-CoV-2 serology test
* Urine pregnancy test (women) Visit 12 - 6 months Final visit Day 180±7 days
* Physical examination (including body weight)
* Vital signs (blood pressure, heart rate, body temperature) measurement
* Blood sample collection for pharmacokinetic analysis
* Blood sample collection for ADA
* Blood sample collection for serum neutralising power test
* Blood sample collection for DIESSE Elisa kit characterisation
* Adverse events monitoring
* Concomitant medications check
* Laboratory analyses: haematology, blood chemistry, urinalysis, coagulation, SARS-CoV-2 serology test
* 12-lead ECG The data documented in this trial and the measured clinical parameters will be presented using classic descriptive statistics for quantitative variables and frequencies for qualitative variables.

A Statistical Analysis Plan will be prepared by CROSS Research S.A. Biometry Unit, approved by the Sponsor and finalised before database lock.

Safety, serum neutralising power, immunogenicity and demography data will be analysed by CROSS Research Biometry Unit using SAS® version 9.3 (TS1M1) or higher (the actual version will be stated in the final report).

Adverse events and serious adverse events (including clinically significant laboratory parameters, vital signs, ECG results and adverse reactions at the injection sites) will be listed by treatment. Number and percentage of subjects with adverse events and serious adverse events will be summarised.

Serum MAD0004J08 concentrations and pharmacokinetic parameters will be analysed using Phoenix WinNonlin® validated version 6.3 or higher (Pharsight Corporation) and SAS® version 9.3 for Windows® or higher. Pharmacokinetics data will be listed and summarised by descriptive statistics. Individual and mean concentration curves will also be generated. ADA concentrations will be summarised by descriptive statistics. Number and percentage of ADA-positive subjects will be listed and summarised by assessment time and overall. Serum neutralising power results will be listed by subject and assessment time-point and summarised by descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent: Signed written informed consent before inclusion in the study
2. Full comprehension: Ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the Investigator and to comply with the requirements of the entire study
3. Sex and age: Healthy men and women, 18 - 55 years old, inclusive
4. Negative SARS-CoV-2 serology test at screening (negative anti-S and anti-N)
5. Negative SARS-CoV-2 qRT-PCR in the 72 h before treatment (test on day -3 or -2 or -1 with result before treatment)
6. Body Mass Index: 18.5-30 kg/m2, inclusive, at screening
7. Vital signs: Systolic blood pressure 90-139 mmHg, diastolic blood pressure 60-90 mmHg, heart rate 50-100 bpm, measured after 5 min at rest in the supine position
8. ECG: Electrocardiogram without clinically significant abnormalities at screening
9. Contraception and fertility: Women of child-bearing potential must be using at least one of the following reliable methods of contraception and confirm to use adequate contraception during the study:

   1. Hormonal oral or implantable or transdermal, or injectable contraceptives for at least 2 months before the screening visit;
   2. A non-hormonal intrauterine device or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide for at least 2 months before the screening visit
   3. A male sexual partner who agrees to use a male condom with spermicide
   4. A sterile sexual partner
   5. A same sex partner Female participants of non-child-bearing potential or in post-menopausal status for at least 1 year will be admitted. For all women, urine pregnancy test result must be negative at screening and day 1

Exclusion Criteria:

1. Physical findings: Clinically significant abnormal physical findings which could interfere with the objectives of the study
2. Allergy: Ascertained or presumptive hypersensitivity to the active principle and/or ingredients of the investigational products; history of anaphylaxis to drugs or allergic reactions likely to be exacerbated by any component of the investigational products in the Investigator's opinion
3. Concomitant medications: Medications, including over the counter (OTC) medications and herbal remedies, for 2 weeks before screening and immunoglobulin or blood products for 6 months before screening (except contraceptives or a single use of paracetamol, aspirin, or combination OTC products containing paracetamol with an antihistamine, or OTC non-steroidal anti-inflammatory drugs (NSAIDs) at a dose equal or lower than that recommended on the package; vitamins and nutritional supplements, if regularly taken before the study, are also allowed)
4. Monoclonal Antibodies (mAb): Previous intake of a mAb within 6 months, or 5 antibody half-life, whichever is longer, before study start
5. Transient acute illness: Acute (time-limited) illness, including fever above 37.5°C on the day before or on the day of the planned treatment; subjects excluded for transient acute illness may be dosed if illness resolves within the screening period or may be rescreened once
6. Diseases: Significant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine, psychiatric or neurological diseases that may interfere with the aim of the study or increase subjects risks; history of malignancy in the last 5 years
7. SARS CoV-2 or COVID-19:

   1. Participants with any confirmed current or previous COVID-19 infection at screening, or at day -1 or day 1
   2. Participant with clinical signs or symptoms consistent with COVID-19, e.g. fever, dry cough, dyspnoea, sore throat, fatigue or confirmed infection by appropriate laboratory test within the last 4 weeks before/at screening or at day -1 or day 1
   3. Any prior intake of investigational or licenced vaccine indicated for the prevention of SARS CoV-2 or COVID-19 or expected intake during follow-up period
   4. Has been reported as a case (confirmed or probable) of COVID-19 from the regional health system
8. Immunodeficiency due to illness, including HIV infection (positivity to anti-HIV-Ab), or due to drugs, including any course of glucocorticoid therapy exceeding 2 weeks of prednisone or equivalent within 6 months before screening.
9. Infections: History of active infection with hepatitis B or C or positive test result for anti-HCV-Ab or HBsAg or anti-HBc-Ab at screening; history of infection with SARS or MERS
10. Laboratory analyses: Abnormal laboratory values that in the opinion of the Investigator are clinically significant
11. Investigative drug studies: Participation in the evaluation of any investigational product for 6 months before this study
12. Blood donation: blood donations for 3 months before the study, during the study and in the 3 months after the end of the study
13. Drug test: positive drug test at screening or day -1
14. Drug, alcohol: history of drug or alcohol abuse within 6 months before screening
15. Pregnancy (women only): positive or missing pregnancy test at screening or day 1; pregnant or lactating women
16. Other: Any condition that might compromise study subject's safety or interfere with the study evaluations or interpretation of subject's safety or study results

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
Severe/serious treatment-emergent adverse events | From Day 1 to Day 8
  Proportion of subjects with severe / serious treatment-emergent adverse events (TEAEs) (including clinically relevant laboratory abnormalities, vital signs, and adverse reactions at the injection site) in the 7 days post-treatment.

SECONDARY OUTCOMES:
Unsolicited and solicited TEAE | From Day 1 to Day 180
  Proportion of subjects with any unsolicited and solicited TEAE (including clinically relevant laboratory abnormalities, vital signs, and adverse reactions at the injection site) up to each assessment time and throughout the study
Peak Plasma Concentration (Cmax) | At each visit from Day 1 to Day 180
  Evaluation of MAD0004J08 serum concentrations and PK parameter Cmax after single dose of 48 mg, 100 mg and 400 mg.
Area under the concentration-time curve from time zero to time t (AUC0-t) | At each visit from Day 1 to Day 180
  Evaluation of MAD0004J08 serum PK parameter (AUC0-t):
  - Area under the concentration-time curve from time zero to time t (AUC0-t) after single dose of 48 mg, 100 mg and 400 mg
Area under the concentration vs. time curve up to infinity (AUC0-∞) | At each visit from Day 1 to Day 180
  Evaluation of MAD0004J08 serum PK parameter AUC0-∞:
  - Area under the concentration vs. time curve up to infinity (AUC0-∞) after single dose of 48 mg, 100 mg and 400 mg
Time to achieve Cmax (tmax) | At each visit from Day 1 to Day 180
  Evaluation of MAD0004J08 serum concentrations and PK parameter tmax after single dose of 48 mg, 100 mg and 400 mg.
Half-life (t1/2) | At each visit from Day 1 to Day 180
  Evaluation of MAD0004J08 serum concentrations and PK parameter t1/2 after single dose of 48 mg, 100 mg and 400 mg.
Distribution volume (Vz/F) | At each visit from Day 1 to Day 180
  Evaluation of MAD0004J08 serum concentrations and PK parameter Vz/F after single dose of 48 mg, 100 mg and 400 mg.
Total body clearance CLt/F | At each visit from Day 1 to Day 180
  Evaluation of MAD0004J08 serum concentrations and PK parameter CLt/F after single dose of 48 mg, 100 mg and 400 mg.
Number ADA positive subjects | At Day 1, Day 8, Week 2, Month 1, Month 4 and Month 6.
  Number and percentage of ADA positive subjects and mean maximum ADA concentration after single dose of 48 mg, 100 mg and 400 mg MAD0004J08
Percentage of ADA positive subjects | At Day 1, Day 8, Week 2, Month 1, Month 4 and Month 6.
  Number and percentage of ADA positive subjects and mean maximum ADA concentration after single dose of 48 mg, 100 mg and 400 mg MAD0004J08
Neutralising power analysis | At Day 1,Day 3, Day 8, Month 1, Month 4 and Month 6.
  Serum neutralising power at baseline, 48 h post-dose, on day 8, at 1 month (day 30±3), 4 months (day 120±4) and 6 months (180±7) after single dose of 48 mg, 100 mg and 400 mg MAD0004J08

OTHER OUTCOMES:
ELISA DIESSE kit characterisation | At Day 1,Day 3, Day 8, Month 1, Month 4 and Month 6.
  Characterisation of DIESSE ELISA kit on serum samples at baseline, 48 h post-dose, on day 8, at 1 month (day 30±3), 4 months (day 120±4) and 6 months (180±7). A blood sample will be used to evaluate if Diesse Kit, developped by Toscana Life Sciences, would be able to detect administered MAD0004J08.
  This kit is not used to monitor study paramethers.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Paolini, Study Director — Toscana Life Sciences Sviluppo s.r.l.
Locations (2):
- Italy (2):
  - Inmi 'L.Spallanzani' - Irccs, Rome, Lazio
  - Crc - Verona, Verona, Veneto

REFERENCES:
- [Derived] Lanini S, Milleri S, Andreano E, Nosari S, Paciello I, Piccini G, Gentili A, Phogat A, Hyseni I, Leonardi M, Torelli A, Montomoli E, Paolini A, Frosini A, Antinori A, Nicastri E, Girardi E, Plazzi MM, Ippolito G, Vaia F, Della Cioppa G, Rappuoli R. Safety and serum distribution of anti-SARS-CoV-2 monoclonal antibody MAD0004J08 after intramuscular injection. Nat Commun. 2022 Apr 27;13(1):2263. doi: 10.1038/s41467-022-29909-x. PMID 35477725
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343